CLINICAL TRIAL: NCT06908330
Title: Increasing Kindergarten Social-Emotional Skills for Positive Long-Term Mental Health: A Pilot Test of the Strengthening Social-Emotional Skills for Relating and Thriving at School (SSTRS) Program
Brief Title: Increasing Kindergarten Social-Emotional Skills for Positive Long-Term Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine C. Pears, Senior Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH138714 (NIH); R34MH138714 (NIH)
Record Dates: First submitted 2025-03-21; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Parenting Behavior; Social Emotional Competence; Internalizing Behavior; Externalizing Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSTRS group (Experimental): These participants will participate in the SSTRS intervention.
  Interventions: Behavioral: Social-emotional Skills for Thriving and Relating at School Program
- Services as Usual (No Intervention): These participants will receive kindergarten programming as usual.

INTERVENTIONS:
Behavioral: Social-emotional Skills for Thriving and Relating at School Program — The SSTRS Program is a developmentally-tailored, school-based preventive intervention focusing on children and their parents at the critical transition to kindergarten to prevent deficits in children's social-emotional skills-which are known transdiagnostic risk factors for a range of mental health problems. Children receive SSTRS programming during their regular school day for eight weeks at the beginning of the school year. Parents receive SSTRS programming via informational videos and virtual parenting groups during the same time period.
  Arms: SSTRS group

SUMMARY:
The goal of this clinical trial is to learn if the Social-emotional Skills for Thriving and Relating at School (SSTRS) Program can help children entering kindergarten and their families. The main questions it aims to answer are: 1) Do children who participate in SSTRS have better social-emotional skills and mental health? and 2) Do parents who participate in SSTRS have more positive parenting skills and involvement in their children's learning?

Researchers will compare the SSTRS Program to the regular kindergarten curriculum without SSTRS to see if being in SSTRS helps children to have better mental health and parents to have better parenting skills.

Kindergarteners will have daily SSTRS lessons in their kindergarten classes for 8 weeks.

Their parents will watch videos and attend group meetings with other parents and answer questions about their own and their children's behaviors and mental health

ELIGIBILITY:
Inclusion Criteria:

* child entering kindergarten in school that is participiating in the study

Exclusion Criteria:

* being in a classroom in which the teacher or EA was previously trained in another closely-related treatment protocol

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Strengths & Difficulties Questionnaire | Parents will complete the measure at baseline, 2 months post-baseline at the end of the intervention and 9 months post-baseline. Teachers will complete the measure at 9 months post-baseline.
  Parent and teacher report on the 25-item measure yields five subscales: Emotional Symptoms Scale (scores range 0-10, high scores indicate more problems), Conduct Problems Scale (scores range 0-10, high scores indicate more problems), Hyperactivity Scale (scores range 0-10, high scores indicate more problems) , Peer Problems Scale (scores range 0-10, high scores indicate more problems), and Prosocial Scale (scores range 0-10, high scores indicate better social skills). A Total Difficulties Score can also be derived by summing all of the scales except the Prosocial Scale resulting in a score raniging from 0 to 40 with higher scores denoting greater difficulties.
Office discipline referrals | These will be collected at 9 months post-baseline.
  These are records of referrals for serious behaviors within the school setting. They are administartive records.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Pears, Ph.D., Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared to the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available no later than 2027. There is no end date.
Access Criteria: Access will be granted according to the procedures for accessing data from the NDA.
URL: https://nda.nih.gov/